CLINICAL TRIAL: NCT03325504
Title: A Multi-centre, Open-label, Randomized, Comparative Clinical Trial of Two Doses of Bone Marrow Autologous MSC+ Biomaterial vs Iliac Crest Autologous Graft, for Bone Healing in Non-union After Long Bone Fractures
Brief Title: A Comparative Study of 2 Doses of BM Autologous H-MSC+Biomaterial vs Iliac Crest AutoGraft for Bone Healing in Non-Union
Acronym: ORTHOUNION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Prof Enrique Gomez-Barrena, Full Professor and Chair of orthopaedic surgery, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHOUNION; 2015-000431-32 (EudraCT Number); EUCTR2015-000431-32-ES (Registry Identifier: International Clinical Trials Registry Plataform)
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Non Union Fracture
Keywords: Non-union; Advanced therapies; Mesenchymal stem cells; Long bone
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hBM-MSCs-Low Dose (Experimental): Autologous Cultured Mesenchymal Stem Cells +Biomaterial (Low Dose): 100x106 cells
  Interventions: Biological: Cultured Mesenchymal Stem Cells
- hBM-MSCs-High Dose (Experimental): Autologous Cultured Mesenchymal Stem Cells+Biomaterial (High Dose): 200x106 cells
  Interventions: Biological: Cultured Mesenchymal Stem Cells
- Autologous iliac crest graft (Active Comparator): Autologous Iliac Crest Grafting
  Interventions: Procedure: Autologous iliac crest graft

INTERVENTIONS:
Biological: Cultured Mesenchymal Stem Cells — Cultured Mesenchymal Stem Cells obtained from expanded bone marrow
  Arms: hBM-MSCs-High Dose; hBM-MSCs-Low Dose
Procedure: Autologous iliac crest graft — Autologous iliac crest grafting
  Arms: Autologous iliac crest graft

SUMMARY:
ORTHOUNION is a multi-centre, open, comparative, randomized, clinical trial with three parallel arms that aims to compare the efficacy of three treatments to enhance bone healing in patients with long bone non-union.

DETAILED DESCRIPTION:
Bone injuries represent an important world medical problem producing significant healthcare and societal expenditure. While most bone injuries are not severe and are capable of healing through bone regeneration by natural callus formation with standard treatments, severe bone injuries may not heal, becoming an important unmet clinical need.

Non-unions, or pseudarthrosis, may occur in 5% to 20% of long-bone fractures that fail to heal properly after more than 6 months, with morbidity, prolonged hospitalization, and increased expenses. The most commonly accepted standard augmentation to procure fracture and non-union healing consists of autologous bone grafting, obtained from the same patient in a different surgical site and transplanted to the reconstruction site. However, autologous bone grafting has some drawbacks (such as persistent pain, scar, late recovery, limited amount of bone, etc) and a limited regeneration efficacy (success rate of about 74%) and high societal cost. Culture-expanded autologous MSCs combined with biphasic calcium phosphate (BCP) biomaterial granules have been claimed as a solid regenerative medicine alternative to autologous bone grafting in non-unions, although current data are limited. In this context, the ORTHOUNION initiative focuses on the opportunity to test the hypothesis of superiority of MSC, the investigational ATMP, versus the currently accepted standard therapy, iliac crest bone autograft to biologically augment surgical treatment of long-bone non-unions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older, both sexes
2. Traumatic isolated closed or open Gustilo I and II, IIIA and IIIB humerus, tibial or femur diaphyseal or metaphysodiaphyseal fracture with a status of atrophic, oligotrophic or normotrophic non-union.
3. Able to understand, accept and sign informed consent
4. Medical health coverage
5. Able to understand and accept the study constraints

Exclusion Criteria:

1. Hypertrophic non-unions
2. Segmental bone loss requiring specific therapy (bone transport, vascularized graft, large structural allograft, megaprosthesis, etc)
3. Unrecovered vascular or neural injury
4. Other fractures causing interference with weight bearing
5. Visceral injuries or diseases interfering with callus formation (severe cranioencephalic trauma, etc.)
6. Active infection of any location and aetiology
7. Surgical contraindication of any cause
8. Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control.
9. Malignant tumour (past history or concurrent disease)(except carcinoma in situ or basalioma in remission)
10. History of bone harvesting on iliac crest contraindicating new iliac crest bone graft harvesting or bone marrow collection
11. Insulin dependent diabetes
12. Any evidence (confirmed by PCR) of active infection with HIV, Hepatitis B or Hepatitis C infection
13. Any evidence of Syphilis
14. Known allergies to products involved in the production process of MSC
15. Corticoid or immunosuppressive therapy more than one week in the three months prior to study inclusion
16. Autoimmune inflammatory disease
17. Current treatment by biphosphonates not stopped three months prior to study inclusion
18. Impossibility to meet at the appointments for the follow up
19. Participation in another therapeutic trial in the previous 3 months
20. Second non-union in case of bilateral or multiple non-unions (only one non-union per patient will be included in the trial)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Bone consolidation | 12 months after treatment
  The percentage of bone consolidation in the comparator treatment arm ( iliac crest autograft) and experimental treatment arm (mesenchymal cells).

SECONDARY OUTCOMES:
Bone consolidation | 6 and 24 months
  To compare bone consolidation between the experimental arms and the comparator
Radiological Bone consolidation | 6, 12 and 24 months
  To compare bone consolidation, using the REBORNE scale, between the experimental arms and the comparator.
  The REBORNE scale is an ad-hoc and validated scale, developed by Gomez-Barrena et al. (article currently under preparation) as a modification of the RUST score (Whelan, 2010; Journal of Trauma). In the REBORNE scale, the presence/absence of radiological consolidation is evaluated on a total of 4 cortices. Score range from 0 (no bone callus visible) to 4 (callus present with same density as cortical). The total score will be recorded.
Level of Pain | 6, 12 and 24 months
  To compare level of pain (by Numeric Rating Scale [NRS]) between the experimental arms and the comparator.
  The NRS is a scale that rates the patient´s pain from 0-10 (0= no pain, 10= worst pain), at the time of the visit.
Complications | 6, 12 and 24 months
  To compare the rate of complications between the experimental arms and the comparator
Health status | 6, 12 and 24 months
  To compare the health status (by using the Short Form-36 Health Questionnaire) between treatment arms.
  The SF-36 questionnaire is a validated, widely used patient-reported health survey which measures their physical and mental health status. It consists of 36 questions organized in 8 dimensions. The total score will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Gomez-Barrena, Prof, Principal Investigator — Universidad Autonoma de Madrid
Locations (19):
- France (5):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Department of Orthopaedic Surgery, Hospital Henri Mondor, Créteil
  - Department of Orthopaedic Surgery, CHU Nantes, Nantes
  - Department of Orthopaedic Surgery Toulouse University Hospital, Toulouse
  - Department of Orthopaedic Surgery, CHU Tours, Tours
- Germany (4):
  - Universitätsklinikum Frankfurt, Department of Trauma, Hand and Reconstructive Surgery, Frankfurt
  - Universitätsklinikum Freiburg, Klinik für Orthopädie und Unfallchirurgie, Freiburg im Breisgau
  - Universitätsklinikum München, Munich
  - Department of Orthopaedic Trauma, University of Ulm, Ulm
- Italy (3):
  - Istituto Ortopedico Rizzoli, SSD Fisiopatologia Ortopedica e Medicina Rigenerativa, Bologna
  - Arienda Spedali Civili di Brescia II Ortopedia e Traumatologia, Brescia
  - Istituto Ortopedico Galeazzi, Chirugia dell´Anca l, Milan
- Spain (7):
  - Hospital U. Puerta de Hierro-Majadahonda, Servicio de Cirugía Ortopédica y Traumatología, Majadahonda, Madrid
  - Hospital Clínica San Carlos, Servicio de Cirugía Ortopédica y Traumatología, Madrid
  - Hospital U. 12 de Octubre, Servicio de Cirugía Ortopédica y Traumatología, Madrid
  - Hospital U. Gregorio Marañon, Servicio de Cirugía Ortopédica y Traumatología, Madrid
  - Hospital U. La Princesa, Servicio de CirugíaOrtopédica y Traumatología, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Servicio de Cirugía Ortopédica y Traumatología "A", Hospital La Paz, Madrid

REFERENCES:
- [Background] Gomez-Barrena E, Padilla-Eguiluz NG, Avendano-Sola C, Payares-Herrera C, Velasco-Iglesias A, Torres F, Rosset P, Gebhard F, Baldini N, Rubio-Suarez JC, Garcia-Rey E, Cordero-Ampuero J, Vaquero-Martin J, Chana F, Marco F, Garcia-Coiradas J, Caba-Dessoux P, de la Cuadra P, Hernigou P, Flouzat-Lachaniette CH, Gouin F, Mainard D, Laffosse JM, Kalbitz M, Marzi I, Sudkamp N, Stockle U, Ciapetti G, Donati DM, Zagra L, Pazzaglia U, Zarattini G, Capanna R, Catani F. A Multicentric, Open-Label, Randomized, Comparative Clinical Trial of Two Different Doses of Expanded hBM-MSCs Plus Biomaterial versus Iliac Crest Autograft, for Bone Healing in Nonunions after Long Bone Fractures: Study Protocol. Stem Cells Int. 2018 Feb 22;2018:6025918. doi: 10.1155/2018/6025918. eCollection 2018. PMID 29535772
- See also: Webpage of the Orthounion Study — http://orthounion.eu